CLINICAL TRIAL: NCT04051281
Title: A Letter From the CMO in England to Reduce Antibiotic Prescribing in General Practice: A Randomized Controlled Trial Comparing Monitoring and Feedback (With and Without Graphs), and Social Norms Feedback (Without and Without a Specific Case Study of Patient Harm)
Brief Title: CMO Letter to Reduce Inappropriate Antibiotic Prescribing Winter 2019/2020
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMO Letter 2019/20
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Prescribing, Off-Label
Keywords: antimicrobial resistance; social norms feedback; behavioural science; feedback and monitoring
MeSH Terms: interventions — College Fraternities and Sororities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Just under target control (No Intervention): Practices whose prescribing in the past year was under the new target but who would exceed the target if they had a 5% increase in prescribing; no letter sent.
- Just under target letter (Experimental): Practices whose prescribing in the past year was under the new target but who would exceed the target if they had a 5% increase in prescribing: receive a letter informing of this.
  Randomization is stratified according to whether their prescribing had increased by > 5% compared to the previous year; those whose prescribing had increased had it mentioned in the letter
  Interventions: Behavioral: Letter
- Over target control (No Intervention): Practices whose prescribing in the past year was above the new target but who were not in the top 20% of prescribers; no letter sent
  * Intervention 1: Letter informing them that their practice's prescribing exceeds the new target (Letter B1)
  * Intervention 2: Letter informing them that their practice's prescribing exceeds the new target with a graph representing prescribing relative to the target (Letter B2)
- Over target letter (Experimental): Practices whose prescribing in the past year was above the new target but who were not in the top 20% of prescribers; receive a letter informing them that their practice's prescribing exceeds the new target (Letter B1)
  Randomization is stratified according to whether their prescribing had increased by > 5% compared to the previous year; those whose prescribing had increased had it mentioned in the letter
  Interventions: Behavioral: Letter
- Over target letter with bar chart (Experimental): Practices whose prescribing in the past year was above the new target but who were not in the top 20% of prescribers; receive a letter informing them that their practice's prescribing exceeds the new target, including a bar chart showing their prescribing compared to the target (Letter B1)
  Randomization is stratified according to whether their prescribing had increased by > 5% compared to the previous year; those whose prescribing had increased had it mentioned in the letter
  Interventions: Behavioral: Letter
- Top 20% feedback letter control (Active Comparator): Targeting practices that are currently in the top 20% of prescribers; letters informing them of the percentile they are on--standard practice--(Letter C1)
  Randomization is stratified according to whether their prescribing had increased by > 5% compared to the previous year; those whose prescribing had increased had it mentioned in the letter
  Interventions: Behavioral: Letter
- Top 20% above target letter (Experimental): Targeting practices that are currently in the top 20% of prescribers; letters informing them that their prescribing exceeds the new target (Letter C2)
  Randomization is stratified according to whether their prescribing had increased by > 5% compared to the previous year; those whose prescribing had increased had it mentioned in the letter.
  Interventions: Behavioral: Letter
- Top 20% feedback letter with specific example of patient harm (Experimental): Targeting practices that are currently in the top 20% of prescribers
  • Control: Current standard practice, a social norms message, that their practice is in the top 20% of prescribers (Letter C1) Targeting practices that are currently in the top 20% of prescribers; letters informing them of the percentile they are on with a specific example of a case of patient harm caused by antimicrobial resistance (Letter C3)
  Randomization is stratified according to whether their prescribing had increased by > 5% compared to the previous year; those whose prescribing had increased had it mentioned in the letter.
  Interventions: Behavioral: Letter

INTERVENTIONS:
Behavioral: Letter — Letters sent to GPs in relevant practices (prescribing data is by practice, so the practice is the unit of randomization)
  Arms: Just under target letter; Over target letter; Over target letter with bar chart; Top 20% above target letter; Top 20% feedback letter control; Top 20% feedback letter with specific example of patient harm

SUMMARY:
This trial aims to reduce inappropriate prescription of antibiotics and broad spectrum antibiotics by general practitioners (GPs) in England. Unnecessary prescriptions are defined as those that do not improve patient health outcomes. The intervention is to send GPs a letter from the Chief Medical Officer (CMO) that gives feedback on their practice's prescribing levels.

There will be three intervention samples:

1. practices whose prescribing in the past year was under the new target of 0.965 items per STAR-PU but who would exceed the target if they had a 5% increase in prescribing; trial compares prescribing of practices whose GPs receive a letter informing them that their practice's prescribing is just under the new target to that of practices that are not sent a letter
2. Practices whose prescribing in the past year was above the new target but who not in the top 20% of prescribers; trial compares prescribing of practices whose GPs receive a letter informing them that their practice's prescribing exceeds the new target to practices who get a letter that includes a graph showing their prescribing relative to the target and to practices that are not sent a letter
3. Practices that are currently in the top 20% of prescribers; trial compares effect on prescribing of a feedback letter with a social norms message (current standard practice for this group) to a letter informing GPs that their practice's prescribing exceeds the new target and to a letter with a social norms message, that includes a specific example of a case of patient harm caused by antimicrobial resistance.

DETAILED DESCRIPTION:
The study will involve three trials, each conducted as non-blinded randomised controlled trial, with GP practices as the unit of randomisation.

Trial 1 Targeting practices whose prescribing in the past year was under the new target but who would exceed the target if they had a 5% increase in prescribing

* Control: No letter
* Intervention: Letter informing them that their practice's prescribing is just under the new target (Letter A) Trial hypothesis: Sending a letter to GPs whose practices are just under the new prescribing target will reduce antibiotic prescribing

Trial 2 Targeting practices whose prescribing in the past year was above the new target but who not in the top 20% of prescribers

* Control: No letter
* Intervention 1: Letter informing them that their practice's prescribing exceeds the new target (Letter B1)
* Intervention 2: Letter informing them that their practice's prescribing exceeds the new target with a graph representing prescribing relative to the target (Letter B2) Hypotheses: (i) Sending a letter to GPs whose practices missed the new prescribing target will reduce their prescribing; (ii) A letter with a graph will be more effective than a letter without a graph.

Trial 3 Targeting practices that are currently in the top 20% of prescribers

* Control: Current standard practice, a social norms message, that their practice is in the top 20% of prescribers (Letter C1)
* Intervention 1: Letter informing them that their practice's prescribing exceeds the new target (Letter C2)
* Intervention 2: Social norms message, that they are in the top 20%, with a specific example of a case of patient harm caused by antimicrobial resistance (Letter C3)

Hypotheses: (i) A letter with a social norms message and a specific example of a case where a patient came to harm will be more effective than a feedback letter without a specific example; (ii) A letter telling GPs that they missed the prescribing target will be no less effective than a letter with social norms feedback

For each letter, there will be two versions, one for practices whose prescribing has increased by > 5% in the previous year, informing them of that their prescribing has increased since the previous year, and one for practices whose prescribing has not been increasing.

The letters will signpost GPs to resources to help address patient demand for inappropriate antibiotic prescribing, recognising that many GPs feel that patients expect antibiotics and that GPs may find it difficult to have the necessary patient conversations, especially within a short consultation. As with previous letters, these letters will advise GPs of actions that they can take to reduce inappropriate prescribing, supporting them to have conversations with patients, and there will be TARGET leaflets enclosed.

Power calculation All trials are powered to detect a 2% reduction in prescribing at a significance level of 0.05 with a power of 80%.

Statistical analysis plan In order to test our hypotheses, the investigators will use a fixed effects panel regression model, with time trends accounting for seasonal effects, to estimate the effect of treatment status on prescribing. The investigators will also run ANCOVAs for each month separately and one covering the whole six months of the trial. Analysis will control for baseline prescribing rates and for whether practices got the version of the letter saying that their prescribing has been increasing.

ELIGIBILITY:
Inclusion Criteria:

• GP practices that prescribed more than 0.919 Antibacterial Items/STAR- PU (5% under the target of 0.965) for the twelve months April 2018 - March 2019

Exclusion Criteria:

• Practices in the 99th percentile of prescribers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2963 (Actual)
Dates: Start 2019-08-31 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Total antibiotic prescribing in September | 1 month
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
Total antibiotic prescribing in October | 2 months
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
Total antibiotic prescribing in November | 3 months
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
Total antibiotic prescribing in December | 4 months
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
Total antibiotic prescribing in January | 5 months
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
Total antibiotic prescribing in February | 6 months
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
Total antibiotic prescribing in from September-February | 6 months
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
Proportion of practices in each group whose prescribing was under the target | 8 months
  Whether antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU) for April 2019-March 2020 is under the NHS target of 0.965 items per STAR-PU

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health England, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Note that the trial will use publicly available prescribing data, so any researcher should be able to access it.